CLINICAL TRIAL: NCT03831191
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of LY3375880 in Adult Subjects With Moderate-to-Severe Atopic Dermatitis: The ADmIRe Study
Brief Title: A Study of LY3375880 in Adults With Moderate-to-Severe Atopic Dermatitis
Acronym: ADmIRe
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for lack of efficacy after an interim analysis was performed
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17104; I9N-MC-FCAB (Other: Eli Lilly and Company); 2018-002401-56 (EudraCT Number)
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2020-06

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 50 mg LY3375880 (Experimental): Induction Period:
  Participants received 50 mg LY3375880 administered SC Q4W.
  Interventions: Drug: LY3375880
- 150 mg LY3375880 (Experimental): Induction Period:
  Participants received 150 mg LY3375880 administered SC Q4W.
  Interventions: Drug: LY3375880
- 600 mg LY3375880 (Experimental): Induction Period:
  Participants received 600 mg LY3375880 administered SC Q4W.
  Interventions: Drug: LY3375880
- Placebo (Placebo Comparator): Induction Period:
  Participants received placebo administered subcutaneously (SC) every 4 weeks (Q4W).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3375880 — Administered SC
  Arms: 150 mg LY3375880; 50 mg LY3375880; 600 mg LY3375880
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug LY3375880 is safe and effective in adults with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have diagnosis of AD >= 12 months according to the American Academy of Dermatology criteria.
* Participants must have moderate to severe AD at screening and randomization.
* Participants must have inadequate response to topical medications within 6 months of screening (or history of intolerance).

Exclusion Criteria:

* Participants must not have concurrent treatment with topical or systemic treatments for AD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (58):
- United States (14):
  - Tien Q. Nguyen, MD inc. DBA First OC Dermatology, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - Quest Dermatology Research, Northridge, California
  - Integrative Skin Science and Research, Sacramento, California
  - Arlington Dermatology, Rolling Meadows, Illinois
  - The South Bend Clinic, South Bend, Indiana
  - Dermatology and Skin Cancer Specialists, Rockville, Maryland
  - ActivMed Practices & Research, Inc, Portsmouth, New Hampshire
  - Piedmont Plastic Surgery and Dermatology, Charlotte, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Hightower Clinical Trial Services, Norman, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Clinical Partners LLC, Johnston, Rhode Island
  - Center for Clinical Studies, Houston, Texas
- Argentina (7):
  - DOM- Centro de Reumatologia, CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Instituto de Neumonología y Dermatología, Ciudad Autonoma Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, Ciudad Autonoma Buenos Aires
  - Parra Dermatología, Mendoza
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Austria (3):
  - Universitätsklinikum Graz, Graz, Styria
  - LKH Feldkirch, Feldkirch, Vorarlberg
  - Sozialmed. Zentrum Ost - Donauspital, Vienna
- The Guenther Dermatology Research Centre, London, Ontario, Canada
- Czechia (2):
  - Clintrial, s.r.o., Prague, Hl. M. Praha
  - Sanatorium Profesora Arenbergera, Prague
- CHU de Nice Hopital de L'Archet, Nice, France
- Germany (2):
  - Dermatologikum Hamburg, Hamburg
  - TFS Trial Form Support GmbH, Hamburg
- Hungary (4):
  - Oroshaza Varosi Onkormanyzat Korhaza, Orosháza, Bekes County
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - UNO Medical Trials Kft., Budapest
  - MedMare Bt, Veszprém
- Italy (3):
  - Policlinico di Tor Vergata, Rome, Lazio
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Polic.Umberto I -Univ. La Sapienza, Roma
- Japan (10):
  - Yasumoto Dermatology Clinic, Chikushino-shi, Fukuoka
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Meiwa Hospital, Nishinomiya, Hyōgo
  - Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Oita University Hospital, Yufu-shi, Oita Prefecture
  - Kume Clinic, Nishi-ku Sakai-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Sumire Dermatology Clinic, Edogawa-ku, Tokyo
  - Matsuda Tomoko Dematological Clinic, Fukuoka
- Mexico (2):
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - Derma Norte del Bajío, S.C., Aguascalientes
- Puerto Rico (5):
  - Office of Dr. Samuel Sanchez PSC, Caguas, PR
  - Office of Dr. Alma M. Cruz, Carolina, PR
  - Ponce School of Medicine CAIMED Center, Ponce, PR
  - GCM Medical Group PSC, San Juan, PR
  - Clinical Research Puerto Rico, Inc., San Juan
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Clinica Universidad De Navarra, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Study of LY3375880 in Adults With Moderate-to-Severe Atopic Dermatitis — https://trials.lillytrialguide.com/en-US/trial/4hXeeEjeZhqtnDW4onAZx3#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Responders are participants who achieved a 50% reduction in the Eczema Area and Severity Index score [EASI-50] response, regardless of whether rescue therapy had been initiated during induction period. Participants did not receive 300 mg because the trial was stopped early.
Groups:
- 50 mg LY3375880: Induction Period:
  Participants received 50 milligrams (mg) LY3375880 administered SC Q4W.
- Placebo Responder to Placebo/300 mg LY3375880: Maintenance Period:
  Participants received placebo administered SC Q4W until loss of response then 300 mg LY3375880 SC Q4W .
  Participants had received placebo SC Q4W during the induction period.
- Placebo Non-Responder to 300 mg LY3375880: Maintenance Period:
  Participants received 300 mg LY3375880 administered SC Q4W.
  Participants had received placebo SC Q4W during the induction period.
- 50 mg Responder to Placebo/50 mg LY3375880: Maintenance Period:
  Participants received placebo administered SC Q4W until loss of response then 50 mg LY3375880 SC Q4W.
  Participants had received 50 mg LY3375880 SC Q4W during the induction period.
- 50 mg LY3375880 Responder to 50 mg LY3375880: Maintenance Period:
  Participants received 50 mg LY3375880 administered SC Q4W.
  Participants had received 50 mg LY3375880 SC Q4W during the induction period.
- 50 mg LY3375880 Non-Responder to 150 mg LY3375880: Maintenance Period:
  Participants received 150 mg LY3375880 administered SC Q4W.
  Participants had received 50 mg LY3375880 SC Q4W during the induction period.
- 150 mg Responder to Placebo/150 mg LY3375880: Maintenance Period:
  Participants received placebo administered SC Q4W until loss of response then 150 mg LY3375880 SC Q4W.
  Participants had received 150 mg LY3375880 SC Q4W during the induction period.
- 150 mg LY3375880 Responder to 150 mg LY3375880: Maintenance Period:
  Participants received 150 mg LY3375880 administered SC Q4W.
  Participants had received 150 mg LY3375880 SC Q4W during the induction period.
- 150 mg LY3375880 Non-Responder to 300 mg LY3375880: Maintenance Period:
  Participants received 300 mg LY3375880 administered SC Q4W.
  Participants had received 150 mg LY3375880 SC Q4W during the induction period.
- 600 mg Responder to Placebo/600 mg LY3375880: Maintenance Period:
  Participants received placebo administered SC Q4W until loss of response then 600 mg LY3375880 SC Q4W.
  Participants had received 600 mg LY3375880 SC Q4W during the induction period.
- 600 mg LY3375880 Responder to 600 mg LY3375880; 600 mg LY3375880 Non-Responder to 600 mg LY3375880: Maintenance Period:
  Participants received 600 mg LY3375880 administered SC Q4W.
  Participants had received 600 mg LY3375880 SC Q4W during the induction period.
Period: Induction Period (16 Weeks)
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880 | Placebo Responder to Placebo/300 mg LY3375880 | Placebo Non-Responder to 300 mg LY3375880 | 50 mg Responder to Placebo/50 mg LY3375880 | 50 mg LY3375880 Responder to 50 mg LY3375880 | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 | 150 mg Responder to Placebo/150 mg LY3375880 | 150 mg LY3375880 Responder to 150 mg LY3375880 | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 | 600 mg Responder to Placebo/600 mg LY3375880 | 600 mg LY3375880 Responder to 600 mg LY3375880 | 600 mg LY3375880 Non-Responder to 600 mg LY3375880
Started | 33 | 35 | 34 | 34 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 33 | 35 | 34 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 10 | 14 | 13 | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 21 | 21 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 12 | 15 | 16 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (36 Weeks)
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880 | Placebo Responder to Placebo/300 mg LY3375880 | Placebo Non-Responder to 300 mg LY3375880 | 50 mg Responder to Placebo/50 mg LY3375880 | 50 mg LY3375880 Responder to 50 mg LY3375880 | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 | 150 mg Responder to Placebo/150 mg LY3375880 | 150 mg LY3375880 Responder to 150 mg LY3375880 | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 | 600 mg Responder to Placebo/600 mg LY3375880 | 600 mg LY3375880 Responder to 600 mg LY3375880 | 600 mg LY3375880 Non-Responder to 600 mg LY3375880
Started | 0 (Participants were assigned to this arm during induction period.) | 0 (Participants were assigned to this arm during induction period.) | 0 (Participants were assigned to this arm during induction period.) | 0 (Participants were assigned to this arm during induction period.) | 4 (Participants were assigned to this arm during maintenance period.) | 5 (Participants were assigned to this arm during maintenance period.) | 2 (Participants were assigned to this arm during maintenance period.) | 4 (Participants were assigned to this arm during maintenance period.) | 8 (Participants were assigned to this arm during maintenance period.) | 1 (Participants were assigned to this arm during maintenance period.) | 4 (Participants were assigned to this arm during maintenance period.) | 8 (Participants were assigned to this arm during maintenance period.) | 1 (Participants were assigned to this arm during maintenance period.) | 1 (Participants were assigned to this arm during maintenance period.) | 9 (Participants were assigned to this arm during maintenance period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 4 | 8 | 1 | 4 | 7 | 1 | 1 | 9
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 4 | 5 | 2 | 4 | 8 | 1 | 4 | 7 | 1 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Post-Treatment Follow-Up Period(8 Weeks)
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880 | Placebo Responder to Placebo/300 mg LY3375880 | Placebo Non-Responder to 300 mg LY3375880 | 50 mg Responder to Placebo/50 mg LY3375880 | 50 mg LY3375880 Responder to 50 mg LY3375880 | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 | 150 mg Responder to Placebo/150 mg LY3375880 | 150 mg LY3375880 Responder to 150 mg LY3375880 | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 | 600 mg Responder to Placebo/600 mg LY3375880 | 600 mg LY3375880 Responder to 600 mg LY3375880 | 600 mg LY3375880 Non-Responder to 600 mg LY3375880
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (No participant entered the post follow-up period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Induction Period:
  Participants received placebo administered SC Q4W.
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880 | Total
Number analyzed (Participants) | 33 | 35 | 34 | 34 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.00 (14.98) | 37.70 (16.00) | 39.50 (13.94) | 36.80 (13.84) | 37.80 (14.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 17 | 14 | 58
  Male | 22 | 19 | 17 | 20 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 9 | 8 | 37
  Not Hispanic or Latino | 12 | 14 | 14 | 16 | 56
  Unknown or Not Reported | 12 | 10 | 11 | 10 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 11 | 14 | 10 | 12 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3 | 6
  White | 19 | 19 | 20 | 19 | 77
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 5 | 3 | 5 | 4 | 17
  Austria | 0 | 4 | 1 | 2 | 7
  Canada | 0 | 0 | 3 | 1 | 4
  France | 2 | 1 | 1 | 0 | 4
  Hungary | 1 | 0 | 3 | 1 | 5
  Italy | 1 | 1 | 1 | 3 | 6
  Japan | 10 | 11 | 10 | 10 | 41
  Spain | 0 | 0 | 3 | 1 | 4
  United States | 14 | 15 | 7 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Validated Investigator's Global Assessment for AD (vIGA-AD) of 0 or 1 With a ≥2 Point Improvement
Description: vIGA-AD measures participants' overall severity of their atopic dermatitis (AD), based on a static, numeric 5 point scale from 0 (clear) to 4 (severe). Higher scores indicate greater severity.The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. Non-responder imputation (NRI) method was used to impute missing data.
Time Frame: Week 16
Population: Induction Period: All randomized participants who completed or discontinued the study prior to study termination by the sponsor.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 21 | 20 | 17 | 21
Percentage of participants | 9.5 [2.7 to 28.9] | 5.0 [0.9 to 23.6] | 5.9 [1.0 to 27.0] | 4.8 [0.8 to 22.7]
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; p = 0.638, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.04 to 6.81]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; p = 0.773, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.05 to 8.76]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; p = 0.671, Regression, Logistic; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.05 to 7.26]

2. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI-75)
Description: EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs - by scoring the extent of disease (percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (erythema, edema/papulation, excoriation, and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head and neck, trunk, upper limbs, and lower limbs). Half scores are allowed. Each body site will have a score that ranges from 0 to 72, and the final EASI score will be obtained by weight-averaging these 4 scores. Hence, the final EASI score will range from 0 to 72 (severe) for each time point. A higher score represented greater disease severity.The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score. Non-responder imputation (NRI) method was used to impute missing data.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 21 | 20 | 17 | 21
Percentage of Participants | 19.0 [7.7 to 40.0] | 15.0 [5.2 to 36.0] | 23.5 [9.6 to 47.3] | 0.0 [0.0 to 15.5]
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; p > 0.999, Fisher Exact; Risk Difference (RD) = -4.0, 95% CI 2-sided [-27.2 to 19.9]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; p > 0.999, Fisher Exact; Risk Difference (RD) = 4.5, 95% CI 2-sided [-20.7 to 30.8]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; p = 0.107, Fisher Exact; Risk Difference (RD) = -19.0, 95% CI 2-sided [-40.0 to 0.2]

3. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD-75)
Description: The SCORAD index uses the rule of nines to assess disease extent (head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; and genitals 1%). It evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss in the last 72 hours on visual analogue scales (VAS) of 0 to 10 where 0 is no itch or sleep loss and 10 is worst imaginable itch or sleep loss. These 3 aspects: extent of disease, disease severity, and subjective symptoms combine to give a score between 0(no disease) and 103 (severe disease). Higher scores indicate greater severity.Non-responder imputation (NRI) method was used to impute missing data.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 21 | 20 | 17 | 21
Percentage of participants | 4.8 [0.8 to 22.7] | 5.0 [0.9 to 23.6] | 0.0 [0.0 to 18.4] | 0.0 [0.0 to 15.5]
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; p > 0.999, Fisher Exact; Risk Difference (RD) = 0.2, 95% CI 2-sided [-18.1 to 19.3]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; p > 0.999, Fisher Exact; Risk Difference (RD) = -4.8, 95% CI 2-sided [-22.7 to 14.1]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; p > 0.999, Fisher Exact; Risk Difference (RD) = -4.8, 95% CI 2-sided [-22.7 to 11.2]

4. Secondary Outcome: Percentage of Participants Achieving vIGA-AD of 0
Description: vIGA-AD measures participants overall severity of their atopic dermatitis (AD), based on a static, numeric 5 point scale from 0 (clear) to 4 (severe). Higher scores indicate greater severity. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification. Non-responder imputation (NRI) method was used to impute missing data.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 21 | 20 | 17 | 21
Percentage of participants | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; Risk Difference (RD) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; Risk Difference (RD) = 0.0, 95% CI 2-sided [0.0 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; Risk Difference (RD) = 0.0, 95% CI 2-sided [0.0 to 0.0]

5. Secondary Outcome: Mean Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis-disease extent and clinical signs-by scoring the extent of disease(percentage of skin affected: 0= 0%;1 =1-9%; 2 =10-29%;3 = 30-49%;4 = 50-69%;5 = 70-89%;6 = 90-100%) and the severity of 4 clinical signs (erythema,edema/papulation,excoriation,and lichenification) each on a scale of 0 to 3 (0 = none, absent; 1 =mild; 2 = moderate; 3=severe) at 4 body sites(head and neck,trunk,upper limbs,and lower limbs).Half scores are allowed.Each body site will have a score that ranges from 0 to 72,and the final EASI score will be obtained by weight-averaging these 4 scores.Hence,the final EASI score will range from 0 to 72(severe) for each time point.Higher scores indicate greater severity.Least Squares Mean(LS Means) were calculated using mixed model repeated measures(MMRM) with treatment,region, baseline disease severity,visit,treatment-by-visit-interaction,baseline and baseline-by-visit-interaction as fixed effects.
Time Frame: Baseline, Week 16
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline EASI value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 6 | 8 | 8 | 9
score on a scale | -11.45 (4.68) | -4.90 (4.30) | -5.89 (4.55) | -7.87 (4.02)
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; p = 0.310, Mixed Models Analysis; Median Difference (Net) = 6.55, 95% CI 2-sided [-6.36 to 19.45]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; p = 0.393, Mixed Models Analysis; Mean Difference (Net) = 5.56, 95% CI 2-sided [-7.50 to 18.63]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; p = 0.564, Mixed Models Analysis; Mean Difference (Net) = 3.59, 95% CI 2-sided [-8.91 to 16.08]

6. Secondary Outcome: Mean Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent (head and neck 9%;upper limbs 9% each;lower limbs 18% each;anterior trunk 18%;back 18%;and genitals 1%).It evaluates 6 clinical characteristics to determine disease severity: (1)erythema,(2)edema/papulation, (3)oozing/crusts,(4) excoriation,(5) lichenification, and (6) dryness on a scale of 0 to 3(0=absence,1=mild,2=moderate,3=severe).The SCORAD index also assesses subjective symptoms of pruritus and sleep loss in the last 72 hours on visual analogue scales(VAS) of 0 to 10 where 0 is no itch or sleep loss and 10 is worst imaginable itch or sleep loss.These 3 aspects: extent of disease,disease severity,and subjective symptoms combine to give a score between 0(no disease) and 103(severe disease).Higher scores indicate greater severity. LS Means were calculated using a MMRM model with treatment,region,baseline disease severity,visit, treatment-by-visit-interaction,baseline and baseline-by-visit-interaction as fixed effects.
Time Frame: Baseline, Week 16
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline SCORAD value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 7 | 8 | 8 | 9
score on a scale | -19.27 (5.92) | -11.66 (5.72) | -16.94 (6.03) | -12.75 (5.3)
Statistical Analysis 1: Comparison: Placebo vs 50 mg LY3375880; Test type: Superiority; p = 0.356, Mixed Models Analysis; Mean Difference (Net) = 7.61, 95% CI 2-sided [-8.82 to 24.05]
Statistical Analysis 2: Comparison: Placebo vs 150 mg LY3375880; Test type: Superiority; p = 0.783, Mixed Models Analysis; Mean Difference (Net) = 2.33, 95% CI 2-sided [-14.64 to 19.30]
Statistical Analysis 3: Comparison: Placebo vs 600 mg LY3375880; Test type: Superiority; p = 0.414, Mixed Models Analysis; Mean Difference (Net) = 6.52, 95% CI 2-sided [-9.40 to 22.43]

7. Secondary Outcome: Percentage of Participants Achieving vIGA-AD of 0 or 1 With a >=2-point Improvement at Week 52
Description: as for outcome 4
Time Frame: Week 52
Population: Maintenance Period: All randomized participants who had a >=2-point improvement at Week 52.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Placebo: Participants received placebo administered subcutaneously (SC) every 4 weeks (Q4W).
- 50 mg LY3375880: Participants received 50 mg LY3375880 administered SC Q4W.
- 150 mg LY3375880: Participants received 150 mg LY3375880 administered SC Q4W.
- 300 mg LY3375880: Participants received 300 mg LY3375880 administered SC Q4W.
- 600 mg LY3375880: Participants received 600 mg LY3375880 administered SC Q4W.
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 300 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 8 | 4 | 12 | 13 | 10
Percentage of participants | 0.0 [0.0 to 32.4] | 0.0 [0.0 to 49.0] | 0.0 [0.0 to 24.2] | 0.0 [0.0 to 22.8] | 0.0 [0.0 to 27.8]

8. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve at a Steady State (AUCτ,ss) of LY3375880
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve at a steady state (AUCτ,ss) of LY3375880. The PK model was fit using all quantifiable concentrations that were collected in the study (i.e., from the induction and maintenance periods).
Time Frame: Induction Period: Pre-dose, Day 0, Day 7, Day 14, Day 28, Day 56, Day 112 Post-dose; Maintenance Period:Predose, Day 168; Day 252, Day 364 Post-dose
Population: All randomized participants who received LY3375880 in induction and maintenance period who had evaluable PK data. Participants did not received 300 mg because the trial was stopped early.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per millilitre (ng*h/mL)
Arm/Group | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880
Number analyzed (Participants) | 35 | 34 | 33
Nanograms*hour per millilitre (ng*h/mL) | 4450 (80.2) | 11200 (41.9) | 49000 (40.5)

ADVERSE EVENTS:
Time Frame: Baseline Up To 45 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly
Groups:
- LY3375880-50mg-Q4W-Post-Treatment Follow-Up Period; LY3375880-150mg-Q4W-Post-Treatment Follow-Up Period; LY3375880-600mg-Q4W-Post-Treatment Follow-Up Period; Placebo-Post-Treatment Follow-Up Period: Follow-up: participants did not receive drug during the follow-up period.
Arm/Group | Placebo | 50 mg LY3375880 | 150 mg LY3375880 | 600 mg LY3375880 | Placebo Responder to Placebo/300 mg LY3375880 | Placebo Non-Responder to 300 mg LY3375880 | 50 mg Responder to Placebo/50 mg LY3375880 | 50 mg LY3375880 Responder to 50 mg LY3375880 | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 | 150 mg Responder to Placebo/150 mg LY3375880 | 150 mg LY3375880 Responder to 150 mg LY3375880 | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 | 600 mg Responder to Placebo/600 mg LY3375880 | 600 mg LY3375880 Responder to 600 mg LY3375880 | 600 mg LY3375880 Non-Responder to 600 mg LY3375880 | LY3375880-50mg-Q4W-Post-Treatment Follow-Up Period | LY3375880-150mg-Q4W-Post-Treatment Follow-Up Period | LY3375880-600mg-Q4W-Post-Treatment Follow-Up Period | Placebo-Post-Treatment Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35 | 0/34 | 0/33 | 0/4 | 0/5 | 0/2 | 0/4 | 0/8 | 0/1 | 0/4 | 0/8 | 0/1 | 0/1 | 0/9 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35 | 0/34 | 2/33 | 0/4 | 1/5 | 0/2 | 0/4 | 0/8 | 0/1 | 0/4 | 0/8 | 0/1 | 0/1 | 0/9 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/33 | 9/35 | 12/34 | 12/33 | 1/4 | 4/5 | 1/2 | 1/4 | 2/8 | 1/1 | 1/4 | 3/8 | 0/1 | 0/1 | 2/9 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | 50 mg LY3375880 (N=35) | 150 mg LY3375880 (N=34) | 600 mg LY3375880 (N=33) | Placebo Responder to Placebo/300 mg LY3375880 (N=4) | Placebo Non-Responder to 300 mg LY3375880 (N=5) | 50 mg Responder to Placebo/50 mg LY3375880 (N=2) | 50 mg LY3375880 Responder to 50 mg LY3375880 (N=4) | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 (N=8) | 150 mg Responder to Placebo/150 mg LY3375880 (N=1) | 150 mg LY3375880 Responder to 150 mg LY3375880 (N=4) | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 (N=8) | 600 mg Responder to Placebo/600 mg LY3375880 (N=1) | 600 mg LY3375880 Responder to 600 mg LY3375880 (N=1) | 600 mg LY3375880 Non-Responder to 600 mg LY3375880 (N=9) | LY3375880-50mg-Q4W-Post-Treatment Follow-Up Period (N=0) | LY3375880-150mg-Q4W-Post-Treatment Follow-Up Period (N=0) | LY3375880-600mg-Q4W-Post-Treatment Follow-Up Period (N=0) | Placebo-Post-Treatment Follow-Up Period (N=0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=33) | 50 mg LY3375880 (N=35) | 150 mg LY3375880 (N=34) | 600 mg LY3375880 (N=33) | Placebo Responder to Placebo/300 mg LY3375880 (N=4) | Placebo Non-Responder to 300 mg LY3375880 (N=5) | 50 mg Responder to Placebo/50 mg LY3375880 (N=2) | 50 mg LY3375880 Responder to 50 mg LY3375880 (N=4) | 50 mg LY3375880 Non-Responder to 150 mg LY3375880 (N=8) | 150 mg Responder to Placebo/150 mg LY3375880 (N=1) | 150 mg LY3375880 Responder to 150 mg LY3375880 (N=4) | 150 mg LY3375880 Non-Responder to 300 mg LY3375880 (N=8) | 600 mg Responder to Placebo/600 mg LY3375880 (N=1) | 600 mg LY3375880 Responder to 600 mg LY3375880 (N=1) | 600 mg LY3375880 Non-Responder to 600 mg LY3375880 (N=9) | LY3375880-50mg-Q4W-Post-Treatment Follow-Up Period (N=0) | LY3375880-150mg-Q4W-Post-Treatment Follow-Up Period (N=0) | LY3375880-600mg-Q4W-Post-Treatment Follow-Up Period (N=0) | Placebo-Post-Treatment Follow-Up Period (N=0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (6) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/11 (0) | 1/16 (1) | 0/17 (0) | 0/13 (0) | 0/2 (0) | 0/2 (0) | 0 (0) | 0/1 (0) | 0/3 (0) | 0/0 (0) | 0/2 (0) | 0/3 (0) | 0/0 (0) | 0 (0) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgenetic alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated for lack of efficacy after an interim analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03831191/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03831191/SAP_001.pdf